CLINICAL TRIAL: NCT01079923
Title: Pilot Pharmacokinetic Study of Daily Versus Monthly High-Dose Cholecalciferol Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Bernard Lee, PharmD, BCPS, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-007602
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Volunteers
Keywords: healthy volunteers; healthy subjects; vitamin D; cholecalciferol; vitamin D3; total vitamin D
MeSH Terms: interventions — Single Person; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single High Dose Supplementation (Active Comparator): Age 18 to 40 years, non-pregnant, non-lactating, female subjects .
  Interventions: Dietary Supplement: Single High Dose Cholecalciferol
- Daily Dose Supplementation (Active Comparator): Age 18 to 40 years, non-pregnant, non-lactating, female subjects.
  Interventions: Dietary Supplement: Daily Dose Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Single High Dose Cholecalciferol — Age 18 to 40 years, non-pregnant, non-lactating, female subjects will receive cholecalciferol 150,000 international units orally once (Bio-tech Pharmacal 50,000 IU capsule, Fayetteville, AR).
  Other Names: Vitamin D3
  Arms: Single High Dose Supplementation
Dietary Supplement: Daily Dose Cholecalciferol — Age 18 to 40 years, non-pregnant, non-lactating, female subjects will receive cholecalciferol 5,000 IU capsule, Fayetteville, AR).
  Other Names: Vitamin D3
  Arms: Daily Dose Supplementation

SUMMARY:
Research has shown that Vitamin D is important in preventing rickets in children, osteomalacia in adults, certain cancers, cardiovascular disease, Type 2 Diabetes, and metabolic syndrome. Data suggests that Vitamin D deficiency is common throughout the world. With increasing medical conditions being linked to Vitamin D deficiency, it is suggested that establishing early normal Vitamin D levels is important to long term health.

There are low quantities of maternal Vitamin D that transfer from blood into breast milk. This places nursing infants at risk of developing low Vitamin D levels, and the American Academy of Pediatrics recommends they receive 400 international units (IU) of Vitamin D daily. If nursing mothers were supplemented with oral Vitamin D, this may produce adequate total Vitamin D in the breast milk for the growing infant to consume. By taking this potential therapeutic approach, this would prevent the burden of administering an oral Vitamin D liquid supplement to an infant.

Recent laboratory technology now allows measurement of total Vitamin D (parent Vitamin D2 plus parent Vitamin D3). The main objective of this pilot study is to compare total Vitamin D levels resulting from daily Vitamin D supplementation of 5,000 international units of cholecalciferol (Vitamin D3) orally for 28 days vs. 150,000 international units of cholecalciferol orally once in healthy, non-pregnant, non-lactating female subjects aged 18 � 40. The research results will be used to help identify an optimal dosing regimen to administer to lactating mothers to hopefully deliver adequate total Vitamin D in nursing infants. This separate study will be conducted at a later date under a subsequent protocol.

Previous research has demonstrated that Vitamin D3 levels become undetectable within 14 days after adult subjects received 100,000 international units of cholecalciferol. The investigators' central hypothesis is that daily dosing of 5,000 international units of cholecalciferol orally will maintain detectable total Vitamin D levels in serum after fourteen days, compared to high-dose 150,000 international units of oral cholecalciferol once.

It is anticipated the aims of this pilot study will yield the following results. First, we, the investigators, hope to determine the resulting Vitamin D blood levels and calculate an appropriate dosing strategy for future research. Next we plan to measure the resulting 25,hydroxyvitamin D levels that correspond with these dosing regimens, since 25,hydroxyvitamin D is the major indicator of Vitamin D status in humans. Lastly, we will measure blood calcium and phosphorus levels to assure these doses of Vitamin D are tolerated by healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* non-pregnant
* non-lactating
* female
* willing to participate in study with adequate compliance and follow-up

Exclusion Criteria:

* Any clinically significant underlying chronic disease states (i.e. diabetes, asthma, seizure disorders, hypo/hyperthyroidism, hypercalcemia, hypophosphatemia, other endocrine disorders, absorption disorders)
* allergy to study medication or its components
* significant travel south of the 35° North latitude in the 28-day study period
* chronic use of steroids, anti-convulsants, or barbiturates
* participation in indoor tanning practices during the 28-day study period

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Vitamin D pharmacokinetics | 28 days
  Characterize the differences in pharmacokinetics of oral Vitamin D3 between two dosing regimens within women of child-bearing age by evaluating any changes in the number of days of detectable total serum Vitamin D and area under the curve (AUC) above baseline.

SECONDARY OUTCOMES:
Vitamin D Supplementation Dosing Regimen | 28 days
  Determine a Vitamin D3 dosing regimen that produces more days of detectable total serum Vitamin D to be used in an additional study examining the quantity of maternal vitamin D that crosses into breast milk for feeding infants.
Vitamin D Supplementation Dosing Regimen Efficacy | 28 days
  Assess differences in change in baseline 25-OH-D between two dosing regimens.
Vitamin D Supplementation Safety | 28 days
  Monitor for any adverse effects of Vitamin D supplementation, specifically hypercalcemia and hypophosphatemia.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard R Lee, PharmD, BCPS, Principal Investigator — Mayo Clinic; Thomas D Thacher, MD, Principal Investigator — Mayo Clinic; Michael E Meekins, PharmD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Holick MF. Vitamin D: importance in the prevention of cancers, type 1 diabetes, heart disease, and osteoporosis. Am J Clin Nutr. 2004 Mar;79(3):362-71. doi: 10.1093/ajcn/79.3.362. PMID 14985208
- [Background] Ford ES, Ajani UA, McGuire LC, Liu S. Concentrations of serum vitamin D and the metabolic syndrome among U.S. adults. Diabetes Care. 2005 May;28(5):1228-30. doi: 10.2337/diacare.28.5.1228. No abstract available. PMID 15855599
- [Background] Foss YJ. Vitamin D deficiency is the cause of common obesity. Med Hypotheses. 2009 Mar;72(3):314-21. doi: 10.1016/j.mehy.2008.10.005. Epub 2008 Dec 2. PMID 19054627
- [Background] Suskind DL. Nutritional deficiencies during normal growth. Pediatr Clin North Am. 2009 Oct;56(5):1035-53. doi: 10.1016/j.pcl.2009.07.004. PMID 19931062
- [Background] Heaney RP, Armas LA, Shary JR, Bell NH, Binkley N, Hollis BW. 25-Hydroxylation of vitamin D3: relation to circulating vitamin D3 under various input conditions. Am J Clin Nutr. 2008 Jun;87(6):1738-42. doi: 10.1093/ajcn/87.6.1738. PMID 18541563
- [Background] Hathcock JN, Shao A, Vieth R, Heaney R. Risk assessment for vitamin D. Am J Clin Nutr. 2007 Jan;85(1):6-18. doi: 10.1093/ajcn/85.1.6. PMID 17209171
- [Background] Mastaglia SR, Mautalen CA, Parisi MS, Oliveri B. Vitamin D2 dose required to rapidly increase 25OHD levels in osteoporotic women. Eur J Clin Nutr. 2006 May;60(5):681-7. doi: 10.1038/sj.ejcn.1602369. PMID 16391587
- [Background] Ilahi M, Armas LA, Heaney RP. Pharmacokinetics of a single, large dose of cholecalciferol. Am J Clin Nutr. 2008 Mar;87(3):688-91. doi: 10.1093/ajcn/87.3.688. PMID 18326608
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Thacher TD, Obadofin MO, O'Brien KO, Abrams SA. The effect of vitamin D2 and vitamin D3 on intestinal calcium absorption in Nigerian children with rickets. J Clin Endocrinol Metab. 2009 Sep;94(9):3314-21. doi: 10.1210/jc.2009-0018. Epub 2009 Jun 30. PMID 19567516
- [Background] Saadi HF, Dawodu A, Afandi B, Zayed R, Benedict S, Nagelkerke N, Hollis BW. Effect of combined maternal and infant vitamin D supplementation on vitamin D status of exclusively breastfed infants. Matern Child Nutr. 2009 Jan;5(1):25-32. doi: 10.1111/j.1740-8709.2008.00145.x. PMID 19161542
- [Background] Armas LA, Hollis BW, Heaney RP. Vitamin D2 is much less effective than vitamin D3 in humans. J Clin Endocrinol Metab. 2004 Nov;89(11):5387-91. doi: 10.1210/jc.2004-0360. PMID 15531486
- [Background] Taylor SN, Wagner CL, Hollis BW. Vitamin D supplementation during lactation to support infant and mother. J Am Coll Nutr. 2008 Dec;27(6):690-701. doi: 10.1080/07315724.2008.10719746. PMID 19155428